CLINICAL TRIAL: NCT04918589
Title: Effects of Tranexamic Acid for Alloplastic Breast Reconstruction: A Randomized Control Trial
Brief Title: Tranexamic Acid for Alloplastic Breast Reconstruction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13104
Record Dates: First submitted 2021-06-04; First posted 2021-06-09 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Hematoma Postoperative; Breast Cancer; Tranexamic Acid
Keywords: Alloplastic Breast Reconstruction
MeSH Terms: conditions — Breast Neoplasms | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT) with 2 arms: the interventional arm (receiving topical TXA) and the control arm (receiving placebo).
  Intervention: Topical application of 3 grams of tranexamic acid (30 mL of 100 mg/mL) diluted in 10 mL of normal saline in the breast.
  Placebo: Topical application of 40 mL of 0.9% normal saline to the breast.
Who Masked: Participant, Care Provider
Masking Description: Patients will be randomized on the REDCap system. Their assignment will be made available to research team member, which will be preparing syringes with either TXA or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic Acid (Experimental): 3 grams of tranexamic acid (30 mL of 100 mg/mL solution) diluted in 10 mL of normal saline
  Interventions: Drug: Tranexamic acid
- Normal Saline (Placebo Comparator): 40 mL topical of 0.9% normal saline
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Tranexamic acid — 3 grams of tranexamic acid (30 mL of 100 mg/mL solution) diluted in 10 mL of normal saline
  Other Names: TXA
  Arms: Tranexamic Acid
Drug: Normal Saline — 40 mL topical of 0.9% normal saline
  Other Names: NS
  Arms: Normal Saline

SUMMARY:
Hematoma is a common complication of alloplastic breast reconstruction. This can lead to pain and discomfort experienced by the patient, in addition to greater use of valuable healthcare resources. Previous studies have shown correlation between the use of tranexamic acid (TXA), an anti-fibrinolytic, and reduced post-surgical bleeding complication events.

In this randomized control trial (RCT) assessing TXA use in alloplastic breast reconstruction, one breast will be randomized to have TXA applied topically, while the other will have normal saline (NS) placebo applied. The primary objective of this prospective blinded randomized control trial study is to determine if the administration of topical TXA in alloplastic breast reconstruction reduces the incidence of surgical site hematoma compared to placebo within 2 weeks following surgery. The results of this study will be used to inform the design of a larger multicentered RCT on TXA in breast surgery.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the use of topical application of tranexamic Acid (TXA) to the surgical wound as a means to decrease hematoma formation compared to placebo in patients undergoing alloplastic breast reconstruction. This project is designed as a single-center RCT to evaluate the effectiveness of topical TXA in this patient population.

If enrolled in this study, patients individual breasts will be randomly assigned to one of two treatment groups for to apply to the wound before it is closed.

One breast will have an intravenous form of TXA applied topically to the surgical site. The other will be have a topical normal saline solution applied to the wound before closure (a placebo).

The patients will have the standard number of drains and postoperative instructions for breast reconstruction. They will follow-up at two weeks time in clinic for assessment, and emergency room visits will be also be evaluated. Standard of care will be practiced with respect to all procedures and visits.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years or older;
* Are undergoing one- or two-stage bilateral alloplastic breast reconstruction immediately after bilateral mastectomy at either Hamilton Health Sciences or St. Joseph's Hospital Hamilton.

Exclusion Criteria:

* Taking therapeutic anticoagulation;
* Taking antiplatelet drugs;
* Pregnant or breast feeding;
* Allergic to TXA;
* Cannot provide informed consent;
* Alloplastic reconstruction is not performed immediately after mastectomy;
* Have a documented coagulopathy or bleeding disorder, acquired disturbances of colour vision, subarachnoid hemorrhage, hematuria, irregular menstrual bleeding, or seizure disorder.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Hematoma | 2 weeks
  Incidence rate of hematoma
Seroma | 2 weeks
  Incidence rate of seroma

SECONDARY OUTCOMES:
Drain output | 24 hours
  Total drain output (mL) at 24 hours
Days with drains | 2 weeks
  Total number of days drains in situ with standard discharge criteria
Reoperation rate | 2 weeks
  Number of repeat operations required for patient related to complication
Reintervention rate | 2 weeks
  Rate of subsequent interventions including aspiration, repeat drain insertion or other
Imaging findings | 2 weeks
  Ultrasound findings of hematoma or seroma, if applicable

CONTACTS AND LOCATIONS:
Overall Officials: Ronen Avram, MD, FRCSC, Principal Investigator — McMaster University
Locations (3):
- Canada (3):
  - St. Joseph's Healthcare, King Campus, Hamilton, Ontario
  - St. Joseph's Healthcare, Charlton Campus, Hamilton, Ontario
  - Juravinski Hospital, Hamilton Health Sciences, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ker K, Edwards P, Perel P, Shakur H, Roberts I. Effect of tranexamic acid on surgical bleeding: systematic review and cumulative meta-analysis. BMJ. 2012 May 17;344:e3054. doi: 10.1136/bmj.e3054. PMID 22611164
- [Background] Wong J, Abrishami A, El Beheiry H, Mahomed NN, Roderick Davey J, Gandhi R, Syed KA, Muhammad Ovais Hasan S, De Silva Y, Chung F. Topical application of tranexamic acid reduces postoperative blood loss in total knee arthroplasty: a randomized, controlled trial. J Bone Joint Surg Am. 2010 Nov 3;92(15):2503-13. doi: 10.2106/JBJS.I.01518. PMID 21048170
- [Background] De Bonis M, Cavaliere F, Alessandrini F, Lapenna E, Santarelli F, Moscato U, Schiavello R, Possati GF. Topical use of tranexamic acid in coronary artery bypass operations: a double-blind, prospective, randomized, placebo-controlled study. J Thorac Cardiovasc Surg. 2000 Mar;119(3):575-80. doi: 10.1016/s0022-5223(00)70139-5. PMID 10694619
- [Background] Ipema HJ, Tanzi MG. Use of topical tranexamic acid or aminocaproic acid to prevent bleeding after major surgical procedures. Ann Pharmacother. 2012 Jan;46(1):97-107. doi: 10.1345/aph.1Q383. Epub 2011 Dec 27. PMID 22202494
- [Background] Gomez-Barrena E, Ortega-Andreu M, Padilla-Eguiluz NG, Perez-Chrzanowska H, Figueredo-Zalve R. Topical intra-articular compared with intravenous tranexamic acid to reduce blood loss in primary total knee replacement: a double-blind, randomized, controlled, noninferiority clinical trial. J Bone Joint Surg Am. 2014 Dec 3;96(23):1937-44. doi: 10.2106/JBJS.N.00060. PMID 25471907
- [Background] Wind TC, Barfield WR, Moskal JT. The effect of tranexamic acid on blood loss and transfusion rate in primary total knee arthroplasty. J Arthroplasty. 2013 Aug;28(7):1080-3. doi: 10.1016/j.arth.2012.11.016. Epub 2013 Mar 28. PMID 23541868
- [Background] Wang H, Shen B, Zeng Y. Comparison of topical versus intravenous tranexamic acid in primary total knee arthroplasty: a meta-analysis of randomized controlled and prospective cohort trials. Knee. 2014 Dec;21(6):987-93. doi: 10.1016/j.knee.2014.09.010. Epub 2014 Oct 23. PMID 25450009
- [Background] Knight H, Banks J, Muchmore J, Ives C, Green M. Examining the use of intraoperative tranexamic acid in oncoplastic breast surgery. Breast J. 2019 Sep;25(5):1047-1049. doi: 10.1111/tbj.13409. Epub 2019 Jun 11. No abstract available. PMID 31187540
- [Background] Pinsolle V, Grinfeder C, Mathoulin-Pelissier S, Faucher A. Complications analysis of 266 immediate breast reconstructions. J Plast Reconstr Aesthet Surg. 2006;59(10):1017-24. doi: 10.1016/j.bjps.2006.03.057. Epub 2006 Jun 5. PMID 16996422
- [Background] Nelson JA, Fischer JP, Grover R, Cleveland E, Erdmann-Sager J, Serletti JM, Wu LC. The impact of anemia on microsurgical breast reconstruction complications and outcomes. Microsurgery. 2014 May;34(4):261-70. doi: 10.1002/micr.22202. Epub 2013 Nov 4. PMID 24436188
- [Background] Megson M. Traumatic subcutaneous haematoma causing skin necrosis. BMJ Case Rep. 2011 Jul 20;2011:bcr0520114273. doi: 10.1136/bcr.05.2011.4273. PMID 22689664
- [Background] Rogoff H, Marquez JE, Ghosh K, Jou C, McAuliffe P, Rathi S, Monroig K, Medrano C, Marmor WA, Ferrier A, Kapadia K, Klein G, Huston TL, Ganz J, Dagum AB, Khan S, Bui D. Clinical Outcomes After Hematoma Development: A Study of 627 Tissue Expander Breast Reconstructions. Ann Plast Surg. 2020 Jul;85(S1 Suppl 1):S63-S67. doi: 10.1097/SAP.0000000000002343. PMID 32243320